CLINICAL TRIAL: NCT01454401
Title: LeucoPatch™ Study. A Multicenter Study on the Effect of LeucoPatch™ in Diabetic Foot Ulcers
Brief Title: LeucoPatch™ Study A Multicenter Study on the Effect of LeucoPatch™ in Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reapplix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-4-2010-090
Record Dates: First submitted 2011-10-14; First posted 2011-10-19 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Weekly LeucoPatch treatment (Other): Weekly treatment of diabetic foot ulcers with LeucoPatch
  Interventions: Device: LeucoPatch treatment

INTERVENTIONS:
Device: LeucoPatch treatment — weekly

SUMMARY:
The LeucoPatch™ study goal is to investigate whether the fully autologous growth factor-containing dressing LeucoPatch™ has a positive effect on healing rates of diabetic foot ulcers. The study seeks to gather data for comparison with previous data from similar wounds (historical controls). By subgrouping of the treated wounds (similar to the historical controls used) an assessment of which of the patient and wound-related factors that might indicate a beneficial effect of LeucoPatch™ is sought.

DETAILED DESCRIPTION:
Summary: Treatment Study

The goal of the LeucoPatch ™ study is to investigate the effect of LeucoPatch ™ in diabetic foot ulcer. LeucoPatch ™ is a biologically active dressings which are made solely by the patient's own blood (autologous). It is produced in the CE (European Conformity) marked LeucoPatch™ Device and contains no additives. In this treatment study up to 75 typical diabetic patients with foot ulcers are included. These wounds are typically chronic and lead to reduced quality of life and ability to work, and extensive treatment costs. Furthermore, these wounds often lead to amputations.The study is a multicenter study in which up to 10 wound clinics are expected to be involved.

The primary endpoint is time to complete healing, the secondary endpoint is change in wound size.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type I or Type II Diabetes
* Age of wounds > 6 weeks
* Wound area <10 cm2
* Wounds: Texas degree ≤ type IIa
* Perfusion status: toe pressure> 30 mmHg, or transcutaneous oxygen measurement (TcPO2)> 30 mmHg on the foot (measured within the last 3 months) or palpable foot pulse (equivalent to> 60 mmHg)
* Diabetes control: HbA1c <12%
* Adequate off-loading (Walker, therapy sandals etc.)
* The patient can adhere to the treatment protocol and is expected to conclude the study
* Written informed consent

Exclusion Criteria:

* Non-Danish or Swedish speaking
* Dementia
* Pregnant or nursing women
* The patient cannot tolerate blood donation
* Hemoglobin : < 6,5 mmol/l or 105 g/l
* Haemophilia, Sickle cell anemia, severe thrombocytopenia, and leukemia or blood dyscrasias.
* Patient on dialysis
* Clinical signs of infection - including osteomyelitis (probe to bone).
* Necrosis of the wound
* 40% change (+/-) in ulcer area in a 2-week run-in period with optimal therapy.
* Blood vessel reconstruction within the last 4 weeks.
* Participation in other clinical wound healing studies in the last 30 days.
* Failure to comply with study protocol in the 2-week run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, MD, Principal Investigator — Dept. of Dermatology D, Bispebjerg Hospital,; Bo Joergensen, MD, Study Director — Dept. of Dermatology D, Bispebjerg Hospital,Denmark; Anna Marie Nielsen, MD, Study Director — University Center for Wound Healing, Odense University Hospital, Denmark; Lise Tarnow, MD,MDSc, Study Director — Steno Diabetes Center, Niels Steensensvej 2, 2820 Gentofte, Denmark; Mariusz Zakrzewski, MD, Study Director — Vascular Center, wound clinic,Kolding Hospital, Skovvangen 2-8,6000 Kolding, Denmark; Niels Ejskjær, MD. PhD, Study Director — Medical Endocrinology, Aarhus University Hospital, 8000 AArhuc C, Denmark; Morten Michelsen, MD, Study Director — Orthopaedic Surgery, Sårcenter. Herlev Hospital, 2730 Herlev, Denmark; Magnus Löndahl, MD. PhD, Study Director — Skane Hospital, Dept Endocrinology, Diabetes Foot Ulcer Clinic, Getingevägen 4, Lund, Sweden; Anders Nilsson, MD, Study Director — Ängelholm Hospital, Diabetes Foot Ulcer Clinic, 262 81 Ängelholm Sweden
Locations (7):
- Denmark (5):
  - Knowledge Center for woundhealing, Bispebjerg Hospital, Copenhagen
  - Steno Diabetes Center, Gentofte Municipality
  - Herlev Hospital, Orthopaedic Surgery Infirmary, Wound Clinic, Herlev
  - Vascular Center, Wound Clinic Kolding Hospital, Kolding
  - University center for woundhealing, Odense Hospital, Odense
- Sweden (2):
  - Ängelholm Hospital, Dept. of Medicine, Diabetic Foot Ulcer Clinic, Ängelholm
  - Skane University Hospital, Dept. of Endocrinology, Diabetes Foot Ulcer Clinic, Lund

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 18-01-2011 (FPI) to 14-01-2013 (LPO)
  Non -ischemic Wagner grade 1 or 2 diabetic foot ulcer (DFU) with a duration of more than 6 weeks and a maximal area of 10 cm2
  Patients with > 40% ulcer area change during a two-week run-in period were excluded.
Pre-assignment Details: 16 patients were excluded during run-in period: >40% ulcer area reduction n=5 HbA1c > 12% n=3 haemoglobin < 9,5% g/dl, n=1 ulcer area > 10 cm2, n=1 amputation n=1 withdrawn consent, n=2 Osteomyelitis n=1 wrongly included n=2
Groups:
- LeucoPatch Treatment of Diabetic Foot Ulcers: Weekly LeucoPatch treatment of diabetic foot ulcers
Period: Overall Study
Arm/Group | LeucoPatch Treatment of Diabetic Foot Ulcers
Started | 44 (ITT)
Completed | 39 (Per Protocol (PP))
Not Completed | 5
Not completed — Death | 1
Not completed — hospitalised | 1
Not completed — osteomyelitis | 2
Not completed — non-adherence | 1

BASELINE CHARACTERISTICS:
Groups:
- LeucoPatch Treatment of Diabetic Foot Ulcers: Weekly treatment
  LeucoPatch device: weekly treatment
Arm/Group | LeucoPatch Treatment of Diabetic Foot Ulcers
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years]
  All | 63 [58 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 35
Diabetes [Number; unit: participants]
  Type 1 | 8
  Type 2 | 36
Body Mass Index (kg/m2) [Median (Inter-Quartile Range); unit: kg/m^2] | 29.7 [25.6 to 32.5]
Presence of neuropathy [Number; unit: participants]
  Yes | 42
  No | 2
Ulcer duration (weeks) [Median (Inter-Quartile Range); unit: weeks] | 35 [16 to 60]
Ulcer area [Median (Inter-Quartile Range); unit: cm^2] | 1.1 [0.5 to 2.9]
Wagner classification [Number; unit: participants] — The Wagner classification is based mainly on wound depth and consists of 6 wound grades. These include: grade 0 (intact skin), grade 1 (superficial ulcer), grade 2 (deep ulcer to tendon, bone, or joint), grade 3 (deep ulcer with abscess or osteomyelitis), grade 4 (forefoot gangrene), and grade 5 (whole foot gangrene).
  participants
    Wagner grade 1 | 19
    Wagner grade 2 | 25
Biochemistry Haemoglobin [Median (Inter-Quartile Range); unit: g/l] | 126 [114 to 139]
Biochemistry [Median (Inter-Quartile Range); unit: 10^9 cells/l]
  Platelets | 262 [225 to 330]
  Leucocytes | 8.0 [6.2 to 10.1]
HbA1c [Median (Inter-Quartile Range); unit: %] | 8.1 [6.2 to 10.1]
HbA1c [Median (Inter-Quartile Range); unit: mmol/mol] | 65 [55 to 79]

OUTCOME MEASURES:

1. Secondary Outcome: Ulcer Healing Within 12 Weeks.
Description: Number of the patients achieved complete epithelialisation at 12 weeks (ITT population) and the percentage respectively in the PP population
Time Frame: 12 weeks
Population: Complete epithelialisation was achieved in 15 patients (34%) in ITT population and 38% in the PP population
Measure: Number; unit: participants
Groups:
- LeucoPatch: LeucoPatch: weekly treatment
Arm/Group | LeucoPatch
Number analyzed (Participants) | 44
participants
  Healed ITT; n=44 | 15
  Healed PP; n=39: number analyzed (Participants) | 39
  Healed PP; n=39 | 15

2. Primary Outcome: Ulcer Healing Within 20 Weeks
Description: Number of the patients achieved complete epithelialization at 20 weeks in the ITT population and in the PP population.
Time Frame: 20 weeks
Population: Number of the patients achieved complete epithelialisation at 20 weeks in the ITT population and in the PP population
Measure: Number; unit: participants
Arm/Group | LeucoPatch
Number analyzed (Participants) | 44
participants
  Healed ITT; n=44 | 23
  Healed PP; n=39: number analyzed (Participants) | 39
  Healed PP; n=39 | 23

ADVERSE EVENTS:
Groups:
- All Patients Consenting to be Enrolled in the Study.: 60 patients were included for a 2 week run-in period. If ulcer area decreased more than 40% during that time the ulcer were deemed "healing" and NOT included for treatment. 16 patients were excluded during the run-in period - 44 were treated. For safety analysis all patients were included
Arm/Group | All Patients Consenting to be Enrolled in the Study.
Serious Adverse Events (participants affected / at risk) | 8/60
Other Adverse Events (participants affected / at risk) | 21/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Consenting to be Enrolled in the Study. (N=60)
SAE not related to Leucopatch treatment (Infections and infestations) | 2 (2)
SAE not related to Leucopatch treatment (Cardiac disorders) | 1 (1)
SAE not related to Leucopatch treatment (Vascular disorders) | 1 (1)
SAE not related to Leucopatch treatment (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SAE not related to Leucopatch treatment (Blood and lymphatic system disorders) | 1 (3)
SAE not related to Leucopatch treatment (Cardiac disorders) | 2 (2)
SAE not related to Leucopatch treatment (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Consenting to be Enrolled in the Study. (N=60)
AE (Infections and infestations) | 1 (1)
AE (Skin and subcutaneous tissue disorders) | 1 (1)
AE (Skin and subcutaneous tissue disorders) | 2 (2)
AE (Investigations) | 2 — Two weeks between treatments
AE (Surgical and medical procedures) | 1 (1)
AE (Blood and lymphatic system disorders) | 1 (2)
AE (Gastrointestinal disorders) | 1 (1)
AE (Renal and urinary disorders) | 1 (1)
AE (Blood and lymphatic system disorders) | 2 (2)
AE (Blood and lymphatic system disorders) | 2 (2)
AE (Skin and subcutaneous tissue disorders) | 1 (1) — Stinging sensation in wound area
AE (Metabolism and nutrition disorders) | 1 (1) — Hypertension medication stop
AE (Renal and urinary disorders) | 1 (1)
AE (General disorders) | 1 (2) — Not taken medication
AE (Injury, poisoning and procedural complications) | 1 (1)
AE (Skin and subcutaneous tissue disorders) | 1 (1)
AE (General disorders) | 1 (3) — Problem blood taking
AE (General disorders) | 1 (1) — Device related problems
AE (Skin and subcutaneous tissue disorders) | 1 (1) — Increase in exudate
AE (Skin and subcutaneous tissue disorders) | 1 (1)
AE (Skin and subcutaneous tissue disorders) | 1 (1) — Blister after footbath
AE (General disorders) | 1 (1)
AE (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No